CLINICAL TRIAL: NCT03237702
Title: Decipher the Biology of Lethal Prostate Cancer - Urine Metabolomics Profiling in Men Receiving Prostate Biopsy and Men With Diagnosed Prostate Cancer Receiving MCS Supplementation
Brief Title: Decipher Lethal Prostate Cancer Biology - Urine Metabolomics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Medical University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Cardinal Tien Hospital (Other); Taipei Medical University Shuang Ho Hospital (Other); Far Eastern Memorial Hospital (Other); Taichung Tzu Chi Hospital (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 201705040MIPB
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Significant Prostate Cancer
Keywords: prostate cancer; prostate biopsy; biomarkers; metabolomics; overtreatment; cancer screening; urine; lycopene; proteomics; urine omics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 1,980 male patients who are planning to have prostate biopsy will be enrolled in the first stage of this study for measuring urine metabolomics. Only the patients who have non-metastatic significant prostate cancer, insignificant prostate cancer, ASAP/PIN, or benign prostate proved by prostate biopsy are enrolled into the second stage in which MCS supplementation will be used for 8 weeks.
  In addition, 20 men and 20 women will be enrolled as a healthy control without any further medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCS arm (Experimental): The participants who will have Multi-Carotenoids for 8 weeks The intervention is Multi-Carotenoids 30 mg for 8 weeks.
  Interventions: Dietary Supplement: Multi-Carotenoids

INTERVENTIONS:
Dietary Supplement: Multi-Carotenoids — All participants in the second stage will receive multi-carotenoids 30 mg qd for 8 weeks.

SUMMARY:
Through a better understanding of the biology of significant (lethal) prostate cancer, we hope to develop new markers/targets from urine metabolomics for more effective screening and prevention of significant prostate cancer. In the meantime, with these new markers we may substantially reduce overtreatment of insignificant PC.

DETAILED DESCRIPTION:
Prostate cancer (PC) afflicts millions of men worldwide. In Taiwan, around 5,000 men are diagnosed as PC while 1,200 men die of the disease each year. However, thousands of Taiwanese men may have been over-treated for their insignificant PCs. The above situations signify the unmet clinical need where effective measures of stratifying risk of PC are lacking. The study is to identify new markers/targets with which to better screen and prevent significant (sPC) or lethal PC (lePC).

This is a prospective, observational and investigational study investigating the role of urine omics studies (metabolomics and proteomics) in subjects who will undergo prostate biopsy or have completed biopsy and/or subsequent MCS supplementation. MCS (or Botreso) is a new patented botanic agent, composed of primarily multi-carotenoids, including lycopene, phytoene, phytofluene, etc. The expected subject number to be enrolled is 620 men and 20 women from NTUH. There will be 3 cohorts: Cohort A (N=990), Cohort B (N=990) and Cohort C (N=40). Cohort A will be the training cohort used to generate the predictive model. Cohort B will be the validation cohort used to validate the newly developed predictive model. Cohort C is the control cohort, including 20 women and 20 men without any signs of cancers.

By risk stratification after biopsy pathology results are available, there will be 5 groups of subjects, including patients with Group 1. mPC: Metastatic prostate cancer Group 2. sPC: Non-metastatic significant prostate cancer (sPC) Group 3. isPC: Non-metastatic insignificant PC (isPC) Group 4. Pre-cancerous lesions: atypical small acinar proliferation (ASAP) or prostatic intraepithelial neoplasia (PIN) Group 5. Non-cancer benign pathology

Based on NCCN risk classification, sPC is defined as the followings: unfavorable intermediate-risk, high/very high-risk, or presence of metastasis. The patients with favorable intermediate-risk prostate cancer will be considered as sPC in the prediction model in the population with long life expectancy.

Biopsy pathology report and clinicopathological parameters will be recorded. In addition, transcriptomics study will be performed. Group specific urine omics profiles will be constructed by comparing the outstanding metabolites between groups. These urine omics profiles are constructed so as to efficiently separate groups of graded risk stratification, especially to predict subjects with mPC (Group 1) or sPC (Group 2). The newly constructed urine omics profiles from Cohort A will be validated against Cohort B of subjects who will undergo biopsy to determine the predictive efficiency of the constructed profiles.

In Cohort A, sPC (Group 2), isPC (Group 3), ASAP/PIN (Group 4) and benign pathology patients (Group 5) will further be invited to take MCS supplementation for 8 weeks after the pathology confirmation. The expected enrollment number is 30 for each of the 4 groups (in total 120). Urine samples will be collected before and after 8 weeks of MCS supplementation for metabolomics and proteomics analysis. The effect of MCS supplementation in modifying urine metabolites will be investigated to determine the potential use of MCS in prostate cancer chemoprevention.

Through a better understanding of the biology of significant (lethal) PC, we hope to develop new markers/targets for more effective screening and prevention of sPC. In the meantime, with these new markers we may substantially reduce overtreatment of insignificant PC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have planned to undergo prostate biopsy or have completed biopsy before 6 weeks.
2. Subjects who are aged between 30 and 100 years men.
3. For subjects who are prostate cancer patients for rebiopsy, the testosterone level should be within normal limit (testosterone >1.5 ng/ml).
4. Subjects who understand the entire study procedures and consent to donate his spot urine (once for 50 ml) and agree with subsequent analyses of his clinical information including biopsy results, treatments and outcomes. (Note: Subjects will be told that the urine metabolomics results will not be revealed to them.)

Exclusion Criteria:

1. Subjects who have other active cancers. However, subjects who have cancers that have been curatively treated and who are disease-free for 3 years or longer are allowed to be enrolled.
2. Subjects who have severe organ function impairment which may significantly alter general cell metabolism determined by the investigators, such as or Cre > 3.0, HbA1c > 9.0%, symptomatic heart failure, or other symptomatic metabolic diseases.
3. Subjects who are receiving or have received systemic therapy, such as chemotherapy, androgen deprivation therapy (ADT), immunotherapy, or targeted therapy within 3 months of the screening.
4. Subjects who have been treated with pelvic radiotherapy within 3 months of the screening.
5. Subjects who have significant infection or inflammation within 8 weeks of the biopsy.
6. Subjects who have pyuria (defined as > 5 WBC/HPF) of urinalysis results within 4 weeks of the biopsy
7. Topical or oral prednisolone equivalent dosage larger 10 mg per day for 14 days or more.
8. The last dose of prednisolone is within 4 weeks of the biopsy.
9. Subjects who have a life expectancy less than 12 months.
10. Subjects who use MCS or found supplementation containing large amount of lycopene in recent 60 days or less. The definition of large amount of lycopene is more than 2 mg per day.

Ages: 30 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change of urine metabolomics | 8 weeks
  Observe the change of metabolomics in urine samples collected before and upon the completeness of MCS supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD PhD, Principal Investigator — Department of Urology, National Taiwan University Hospital
Locations (1):
- Department of Urology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No